CLINICAL TRIAL: NCT03633292
Title: Aloe Vera and Chlorhexidine as Preventive Oral Antiseptics Against the Appearance of Traumatic Oral Ulcers in Patients With Fixed Orthodontics: a Randomized Clinical Trial
Brief Title: Aloe Vera and Chlorhexidine Against Traumatic Oral Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Alfonso X El Sabio University (Other)
Responsible Party: Principal Investigator, Mario Pérez Sayáns, Principal investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RCT-04-16
Record Dates: First submitted 2018-06-25; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Oral Ulcer
MeSH Terms: conditions — Oral Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clorhexidine (Active Comparator): - Clorhexidine Gel (LACER®, Barcelona, Spain) 0.12%, application 2 times / days for 1 month. The gel will be applied two times/day each 12 hours to the gingiva and mucosa.
  Interventions: Drug: Antiseptic clorhexidine gel (Lacer, Barcelona, Spain)
- Aloe Vera (Experimental): - 80% Aloe vera gel, application 2 times / day for 1 month
  Master formula of 80% aloe vera gel Aloe Vera extract, obtained from the central part of the caudal leaves of plants with more than 8 years of life, eliminating its bark. Formulated with carbopol, hydrophilic crosslinked polymer of acrylic acid and vitamin C. The mixture is presented in containers that serve as a container for preparation and will be dispensed in the canister format with applicator tube.
  Interventions: Drug: Master formula of aloe vera gel 80%

INTERVENTIONS:
Drug: Antiseptic clorhexidine gel (Lacer, Barcelona, Spain) — Together with the dispensing container, the dosing and dosage of the gel in research will be attached, with the description of the pharmaceutical form, packaging and labeling of the product. Packages with 8 ml of the gel under investigation, sufficient treatment for 1 month of applications. Posology: After tooth brushing, apply a small amount of gel on the fingertip of a freshly washed finger and spread it over the gum, doing a gentle massage, for 15 ", 2 times a day after proper oral hygiene and it is recommended not to ingest no liquid or food until after half an hour of use.
  Arms: Clorhexidine
Drug: Master formula of aloe vera gel 80% — Blindly and in the same container as chlorhexidine, patients will be instructed to apply aloe vera gel on the gums and mucous membranes once the orthodontic appliances have been cemented
  Arms: Aloe Vera

SUMMARY:
The development of gingivitis in patients during orthodontic treatment is widely known, with the characteristic response of gingival inflammation and hyperplasia and traumatic rashes or ulcerations of the oral mucosa derived from the treatment. The use of chemical agents such as CHX, although it has proven to be useful in these patients, but has the disadvantage of having side effects such as staining, even restricting its use during treatment.

The objective of this study was to determine the efficacy of Aloe vera gel at 80% compared to 0.12% Chlorhexidine gel to alleviate the effects derived from any orthodontic treatment, such as gingival inflammation and hyperplasia and friction or ulcerations. of traumatic oral mucosa-derived from treatment in patients after cementation with metal brackets in the two arches. A total of 140 patients between the ages of 10 and 55 who were randomized and assigned in the two study groups treated with Aloe vera gel versus the conventional Chlorhexidine gel with a sample of 70 subjects in each group participated.

The index of gingival inflammation, plaque index, as well as the simplified hemorrhage index, were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have just begun orthodontic treatment after bracket cementation.
* Be willing and have signed the informed consent.
* Presence of cemented metal brackets throughout the upper and lower arches.
* Presence of good oral health: dental, periodontal and soft tissue

Exclusion Criteria:

* Allergic or who have suffered adverse reactions to Chlorhexidine or Aloe Vera.
* Pregnant, since they are not claimants of fixed multibrackets appliances.
* Presence of auxiliary extraoral appliances during the treatment that may cause additional injuries.
* Under 11 years old.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of traumatic oral ulcers | 30 days
  The patient will attend his scheduled appointment for bracket cementation. Before cementing, we will complete the clinical history (frequency of brushing, smoker or non-smoker, age, sex) aided by intraoral photographs, always collected in the same order according to protocol and by the same researcher. After the cementation, the patient will be included in the study in a random way in the corresponding group. One month after cementing and coinciding with the periodic visit of the patient, the presence / absence of friction or traumatic ulcers will be evaluated.

SECONDARY OUTCOMES:
Prevalence of gingival inflammation | 30 days
  One month after cementing and coinciding with the periodic visit of the patient, the presence / absence gingival inflammation through the gingival inflammation index will be evaluated.
  0 = Normal gingiva, absence of inflammation, no change in color, no bleeding.
  1 = slight inflammation, slight change in color, small alteration of the surface, no hemorrhage. 2 = Moderate inflammation, redness, edema and hemorrhage on probing and pressure. 3 = Strong inflammation, intense redness, edema, tendency to hemorrhages, eventually ulceration. It is interpreted as follows: Sum of the degree of each face / No. of faces observed 0.0-1.0 = incipient gingivitis 1.1-2.0 = Moderate gingivitis 2,1-3,0 = Severe gingivitis
Prevalence of gingival bleeding | 30 days
  One month after cementing and coinciding with the periodic visit of the patient, the presence / absence of gingival bleeding through the gingival index or Simplified haemorrhage index (DHI). It is taken on four sides of the tooth, distal, vestibular, mesial and palatal. The average of the four measurements will be the value of that patient. Periodontal probe will be used. 0 = absence of hemorrhage; 1 = presence of haemorrhage.

OTHER OUTCOMES:
Security and tolerability - number of participants with treatment related adverse events as assessed by CTCAE v4.0 | 30 days
  The study subject is obliged to communicate, by telephone or personally, any type of symptom: redness (erythema), thickening (edema) and peeling (ulcer) occurred after application of the products under study, and will must immediately interrupt the use of it, registering the adverse effects and number of participants with treatment related adverse events as assessed by CTCAE v4.0 and using as a rescue product for the treatment of contact mucositis and antiallergic drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Pérez Sayáns, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided